CLINICAL TRIAL: NCT03209661
Title: Vascular Effects of a Single Bout of Electronic Cigarette Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2016-04-0115
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Arterial Stiffness
Keywords: vascular function
MeSH Terms: interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Subjects will be asked to inhale one of three mediums; 5.4% NBV e-ciggarette, 0% NBV cigarette, and sham menthol inhaler (no vapor). Baseline measurements will be conducted upon arrival and followed immediately post inhalation, 1-hour post, and finally 2-hours post. All trials will require a minimum of 48 hours washout.
Who Masked: Participant
Masking Description: E-cigarettes being utilized are of the same brand and design. Additionally, the device will be covered by a sheath to ensure labeling is not visible to the subject.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- E-Cigarette 5.4% NBV (Active Comparator): Subjects will be asked to inhale an E-Cigarette with 5.4% NBV for 6 min.
  Interventions: Drug: E-cigarette
- E-Cigarette 0% NBV (Placebo Comparator): Subjects will be asked to inhale an E-Cigarette with 0% NBV for 6 min.
  Interventions: Drug: Nicotine 0%
- Menthol Inhaler (Placebo Comparator): Subjects will be asked to inhale a sham methole inhaler (that looks identical in looks to E-cigarette) for 6 minutes. This arm is to control for a potential effect of menthole.
  Interventions: Drug: Menthol Inhalant Product

INTERVENTIONS:
Drug: E-cigarette — E-Cigarette containing 5.4% nicotine will be administered to determine the effects on vascular function.
  Other Names: Nicotine 5.4%
  Arms: E-Cigarette 5.4% NBV
Drug: Nicotine 0% — E-Cigarette containing 0% nicotine will be administered to determine the effects on vascular function.
  Other Names: Placebo
  Arms: E-Cigarette 0% NBV
Drug: Menthol Inhalant Product — Menthol inhaler will be administered to determine the effects on vascular function.
  Other Names: Placebo
  Arms: Menthol Inhaler

SUMMARY:
Investigating the acute effects of a single use E-Cigarette upon vascular health.

DETAILED DESCRIPTION:
Subjects will inhale e-cigarettes of 5.4%, 0%, and sham menthol inhaler to determine the effects upon to measures of vascular health. These measures will include Cardio-Ankle Vascular Index and Flow Mediated Dilation.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy, with no cardiovascular or metabolic diseases. Additionally, is not a frequent smoker of any kind.

Exclusion Criteria:

* Cardiovascular or Metabolic Diseases and/or regular smoker.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in arterial stiffness and endothelial function with e-cigarette use. | Immediately Post, 1 hour, and 2 hour.
  Arterial stiffness and endothelial function are two of the subclinical markers of vascular dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Tanaka, Phd, Principal Investigator — University of Texas
Locations (1):
- Cardiovascular Aging Research Lab at UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cossio R, Cerra ZA, Tanaka H. Vascular effects of a single bout of electronic cigarette use. Clin Exp Pharmacol Physiol. 2020 Jan;47(1):3-6. doi: 10.1111/1440-1681.13180. Epub 2019 Oct 7. PMID 31531991